CLINICAL TRIAL: NCT05280171
Title: Impact of Teach Back of Discharge Information in Term of Patient Recall of Information and Patient Engagement in Self-care Among Chronic Liver Disease Patients Admitted in Selected Wards of ILBS, New Delhi
Brief Title: Impact of Teach Back of Discharge Information in Term of Patient Recall of Information and Patient Engagement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ILBS-TBDIRPE-101
Record Dates: First submitted 2021-12-29; First posted 2022-03-15 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-01

CONDITIONS: Patient Engagement
Keywords: Teach Back; Recall of Discharge Information; Patient Engagement in self care; Health Literacy; Chronic Liver Disease
MeSH Terms: conditions — Patient Participation | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teach back (Experimental): Discharge information was explained by the principal investigator. It includes pictographs teach back regarding medication, exercise, diet and follow-up was given and they were asked teach back.
  Interventions: Other: Teach back
- Standard of Care (Active Comparator): Discharge information as per the standard existing routine. Than assessed the recall and patient engagement of CLD patients in general ward regarding discharge instructions by structure questionnaires for patients recall, and PAM for patient's
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Teach back — Discharge information was explained by the principal investigator. On the day of discharge, pictographs teach back regarding medication, exercise, diet and follow-up was given and they were asked teach back.
  Teach back is a approach which is used in cognitive psychology experiments describing repeating short sequences of information helps to improve repeat back of information. This teach back technique is recommended as a universal precaution by the agency for healthcare research and quality and the national quality forum.
  Arms: Teach back
Other: Standard of care — Standard of care
  Arms: Standard of Care

SUMMARY:
Impact of Teach Back of Discharge Information in term of patient Recall of Information and patient Engagement in self-care among Chronic Liver Disease patients admitted in selected wards of ILBS, New Delhi

Primary objectives

1. To evaluate the impact of teach back on patient recall of discharge information among Chronic Liver Disease patients.
2. To evaluate the impact of teach back on engagement in self care among Chronic Liver Disease patients.

Secondary objectives

1. To find the association of health literacy with patient recall in experimental group after discharge information.
2. To find the association of health literacy with patient engagement in experimental group after discharge information.
3. To find the association of patient recall with selected demographic and clinical variable in experimental group after discharge information.
4. To find the association of engagement in self-care with selected demographic and clinical variable in experimental group after discharge information.

Assumptions The current study is conceptualized on the basis of the following assumptions

1. It is assumed that the patients health information need to be focused on individual needs to improve their health literacy (Yen&Leasure,2019).
2. It is assumed that teach back method will improve patient's immediate and short term recall of discharge information(Mahajan et al,2020).
3. It is assumed that teach back will support self management and promote health outcome(Yen & Leasure, 2019).

DETAILED DESCRIPTION:
Aim of the study This study is aimed to assess the impact of teach back on Chronic Liver Disease patients recall of discharge information and patient's engagement.

To evaluate the efficacy of teach-back in improving comprehension and engagement in self care at the time of discharge.

Problem statement A quasi experimental study to assess the impact of Teach Back of Discharge Information in terms of patient Recall of information and patient Engagement in self care among Chronic Liver Disease patients admitted in selected wards of ILBS New Delhi.

Assess

Operational Definitions

It means to evaluate and estimate the nature, ability or quality of something. In this study, assess refers to evaluate and estimate, the nature or ability of the patient

recall and engagement regarding discharge information among Chronic Liver Disease patients.

Impact The term impact describes all the changes which are expected to happen due to the implementation and application of a given policy option/intervention.

In this study, impact refers to improved patients recall and engagement in self care with the use of teach back of discharge information.

Teach Back Teach-back is a method of ensuring that the teaching is effective by asking for the learner to teach it back in his or her own words.

Teach back is a communication confirmation method used by Researcher to provide information about their diagnosis ,treatment ,medication, risk of treatment, during discharge, then patients will be clearly describe the information provided by researcher. The researcher will clarify the information as needed in Chronic Liver Disease.

Teach back is an evidence based technique to verify not patient recall ,but also their understanding by asking them to repeat the given discharge information in their own words.

Teach back is an efficient and non time consuming method to improve patients, immediate and short term recall and comprehension of the discharge information

Recall It means remembrance of what has been learned or experienced. In this study, it refers to remembrance of discharge information related to treatment, follow up, and self care of Chronic Liver Disease patients. It is measured by structured recall inventory and each item categorized in complete comprehension>90%, partial 90-65%,minimal 65-40%, none<40 Patient Engagement Patient engagement is defined as a concept that combines a patient's Recall, skills, ability and willingness to manage his/her own health and care with interventions. It increases patient activation and promote positive patient behavior.

In this study refers to patient's Recall, skill, ability and willingness to manage her/ his own health include self-care, to increase activation and promote positive patient behavior. It measured by a 22 item patient activation measure scale and the score are categorized as level 1:<47 not believing activation is important, level 2: 47-55 a lack of Recall and confidence to take action, level 3: 55-67 beginning to take action, level 4:>67 taking action.

Discharge Information Discharge information means documented information relevant to a patient's medical condition or behavioral health issue provided by a health care institution to the patient or the patient's representative at the time of the patient's discharge.

In this study it refers to documented information including patient's treatment,(medical and self care),follow up consultations, and return precautions provided by a health care institution to the Chronic Liver Disease patients at the time of patient's discharge.

Chronic Liver Disease(CLD) Chronic liver disease is a progressive deterioration of liver functions for more than six months, which includes synthesis of clotting factors, other proteins, detoxification of harmful products of metabolism and excretion of bile. Chronic Liver Disease is a continuous process of inflammation, destruction, and regeneration of liver parenchyma, which leads to fibrosis and cirrhosis.

In this study, Chronic liver disease is a progressive deterioration due to inflammation, destruction leading to fibrosis and cirrhosis of liver functions for more than six months. Chronic Liver Disease is diagnosed by the physician and admitted in the selected ward of ILBS for treatment.

Variable of the study Assumptions The current study is conceptualized on the basis of the following assumptions

1. It is assumed that the patients health information need to be focused on individual needs to improve their health literacy (Yen&Leasure,2019).
2. It is assumed that teach back method will improve patient's immediate and short term recall of discharge information(Mahajan et al,2020).
3. It is assumed that teach back will support self management and promote health outcome(Yen &Leasure, 2019).

   Conceptual Framework The present study is based on Iowa Model of Evidence-Based Practice to assess the impact of teach back on patient recall of discharge information and patient engagement among patients with chronic liver disease admitted at ILBS, New Delhi.

   Delimitation of the study The study is delimitation to;

   • The patients with chronic liver disease admitted in general ward of ILBS New Delhi.

   Material and Methods Research Approach Quantitative research approach Research Design: Quasi experimental research design Two group post test only design

   The symbols used means: R:Randomization allocation E:Experimental group C:Comparison group X:Teach back of discharge information, O:Recall and patients' engagement of discharge patients.

   INTERVENTION:

   Teach back is a approach which is used in cognitive psychology experiments describing repeating short sequences of information helps to improve repeat back of information. This teach back technique is recommended as a universal precaution by the agency for healthcare research and quality and the national quality forum.

   Need of teach back:

   Teach back is an important issue for the recommendation , which relates to the time this may be take relative to standard instruction.

   Teach back would likely result in increased nurse time spent in the room at the time of discharge discussing and answering remaining questions.

   Therefore in the current study teach back method is undertaken on the basis of broad literature review find out that teach back are better advanced as a universal precaution or in a more a targeted intervention for patient.

   Setting of the study The study will be conducted in General Ward of ILBS, New Delhi

   Population Target population: Chronic Liver Disease patients Accessible population: Chronic Liver Disease patients in General Ward of ILBS, New Delhi

   Sample Technique Random allocation into experimental and control group.

   Sample Size The sample size for the present study was estimated based on previous research study done on patient 's recall of discharge information regarding chronic liver disease and patient engagement. For this purpose, the literature was reviewed and the study by Mahajan et al.,(2020) was chosen. Assuming the baseline values were same, after the intervention the mean recall of discharge information in experimental group was3.95 ± 0.15 and in comparison group was 3.72 ± 0.4.based on this study ,the sample size was calculated with alpha 5% and power 80 percent using the formula.

   According a total of 54 patients were required to be included in the study,27 in experimental group and 27 in comparison group.

   In anticipation of sample dropout, it was decided to round up the total to 60 patients (30 enrolled in each group) from among those who meet the sample selection criteria.

   Sampling criteria

   Tool for data collection

   There are 4 tools used in this study.

   There are given below:

   Tool-1 Demographic Variables Tool-2 Recall inventory Tool-3Patient Activation Measure (PEM-22) Tool-4 All aspects of health literacy scale (AAHLS)

   Data analysis method Descriptive statistics - Descriptive analysis will be used to calculate mean, percentage distribution and standard deviation, through tabulation and graphic presentation.

   Inferential statistics- Chi square test, independent t-test will be used to measure the relationship between two or more variables (demographic and clinical variable)

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease -

  * Admitted in general ward of ILBS New, Delhi
  * Within the age group 18-65 year
  * Willing to participate.
  * Can understand Hindi or English.

Exclusion Criteria:

* Patients with chronic liver disease -

  * Diagnosis of altered mental status.
  * On hospice care
  * On leaving against medical advice.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Impact of teach back on patient engagement in self care | up to 5 weeks
  Patient engagement in self-care was assessed by the patient activation measure scale of the chronic liver disease patient. It consists of 22 items with minimum 0 and maximum 22 score and whether higher scores mean a better outcome.
Impact of teach back on patient recall of the discharge information | up to 5 weeks
  Assessment using recall inventory consist of 28 items with minimum 0 and maximum 28 score and higher scores mean a better outcome and was assessed by the recall of discharge information that includes medication, diet, exercise and follow-up of chronic liver disease patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sheetal Ms Chhikara, Nursing, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Sheetal Chhikara, New Delhi, National Capital Territory of Delhi, India